CLINICAL TRIAL: NCT02498769
Title: Temporary Autonomic Blockade to Prevent Atrial Fibrillation After Cardiac Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joseph Mathew, M.D. (Other)
Collaborators: Foundation for Anesthesia Education and Research (Other); American Heart Association (Other)
Responsible Party: Sponsor-Investigator, Joseph Mathew, M.D., Jerry Reves, MD, Professor of Cardiac Anesthesiology and Chairman, Department of Anesthesiology, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00061607
Record Dates: First submitted 2015-07-08; First posted 2015-07-15 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation
Keywords: Cardiac Surgery; Postoperative Complications; Autonomic Nerve Block
MeSH Terms: conditions — Atrial Fibrillation; Postoperative Complications | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epicardial Botulinum (Experimental): After instituting cardiopulmonary bypass (CPB), botulinum toxin injections will be performed by the surgeon as follows: Using a standard sterile insulin syringe with a 27g needle, surgeons will inject each of the epicardial fat pads with 50U (1mL) of botulinum toxin (OnabotulinumtoxinA, Botox®). After completion of surgery and separation from CPB, patients will proceed along the institutional Cardiac Surgical Caremap. All patients will be monitored with continuous ECG (telemetry) until hospital discharge. POAF will be diagnosed by telemetry or 12-lead ECG, and will be defined as new-onset if it occurs postoperatively at any time before hospital discharge.
  Interventions: Drug: Botulinum Toxin Type A
- Epicardial Placebo (Placebo Comparator): After instituting cardiopulmonary bypass (CPB), placebo (normal saline) injections will be performed by the surgeon as follows: Using a standard sterile insulin syringe with a 27g needle, surgeons will inject each of the epicardial fat pads with 1mL of normal saline. After completion of surgery and separation from CPB, patients will proceed along the institutional Cardiac Surgical Caremap. All patients will be monitored with continuous ECG (telemetry) until hospital discharge. POAF will be diagnosed by telemetry or 12-lead ECG, and will be defined as new-onset if it occurs postoperatively at any time before hospital discharge.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum Toxin Type A — The botulinum toxin will be injected into epicardial fat pads shortly after cardiopulmonary bypass is initiated.
  Other Names: Botox; Onabotulinumtoxin A
  Arms: Epicardial Botulinum
Drug: Placebo
  Other Names: normal saline
  Arms: Epicardial Placebo

SUMMARY:
In this study, the investigators aim to determine whether injecting botulinum toxin into epicardial fat pads is efficacious and safe for decreasing postoperative atrial fibrillation (POAF) after cardiac surgery. The investigators will test the hypothesis that botulinum toxin injected into the epicardial fat pads reduces POAF and length of stay (LOS) without increasing adverse events. This will be a prospective randomized trial of 130 patients undergoing coronary artery bypass graft (CABG), valve surgery or CABG + valve surgery with cardiopulmonary bypass. Patients will be randomized to receive either botulinum toxin (50 units per fat pad, n=65) or normal saline/placebo (1 mL per fat pad, n=65) injected into epicardial fat pads. All patients will receive standardized anesthetic, surgical, and post-surgical care. The primary outcome in this study will be time to occurrence of in-hospital POAF. Based on previous work and a pilot trial showing a pronounced reduction (relative risk reduction 77%) in POAF after injecting botulinum into the epicardial fat pads, the investigators anticipate a significant reduction in the risk for POAF with epicardial botulinum in this cohort, which includes valve surgery patients.

DETAILED DESCRIPTION:
Purpose of the study: A pilot study to determine whether injecting botulinum toxin into epicardial fat pads is efficacious and safe for decreasing postoperative atrial fibrillation (POAF) after cardiac surgery

Hypothesis to be tested: Botulinum toxin injected into the epicardial fat pads reduces POAF.

Design and Procedures: This will be a prospective randomized pilot trial of 130 patients undergoing coronary artery bypass graft (CABG), valve surgery or CABG + valve surgery via median sternotomy with cardiopulmonary bypass. Patients <50 years of age, with chronic atrial fibrillation, prior cardiac surgery, EF<25%, preoperative inotropic support, hepatic or renal failure, known sensitivity to botulinum toxin, debilitating neuromuscular disease, or those with a history of atrioventricular block will be excluded from the study. Prior to surgery, all patients will have baseline Mini-Mental State Examination (MMSE) and blood sampling from an indwelling arterial line or venipuncture for measurement of inflammatory and genomic markers. Half of the patients will be randomized to receive injection of epicardial botulinum toxin in addition to standard of care, as described below. The other half will receive epicardial injection of normal saline.

Institution of cardiopulmonary bypass will be performed according to the routine surgical protocol. After instituting CPB, botulinum toxin (or normal saline) injections will be performed by the surgeon. This dose was selected given the prior report of its effectiveness in preventing POAF after cardiac surgery in a small pilot study.(Pokushalov et al., 2014) After completion of surgery and separation from CPB, patients will proceed along the institutional Cardiac Surgical Caremap. All patients will be monitored with continuous ECG (telemetry) until hospital discharge. POAF will be diagnosed by telemetry or 12-lead ECG, and will be defined as new-onset if it occurs postoperatively at any time before hospital discharge. POAF, if it occurs, will be treated as per routine of care. POAF will be defined as any detectable atrial fibrillation before discharge that lasts >30 seconds. On postoperative day (POD) 4, a member of the study team will visit each patient to administer the MMSE and capture a 5-minute ECG with a Holter monitor. In addition, patients will be contacted monthly for 4 months and at one year after surgery for follow up, and medical records will be reviewed for evidence of readmissions, arrhythmias, or other adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiac surgery with cardiopulmonary bypass via median sternotomy
* coronary artery bypass graft (CABG)
* valve surgery
* CABG + valve surgery

Exclusion Criteria:

* < 50years of age
* > 90years of age
* chronic AF or AF at the time of screening
* preoperative heart block (second degree or greater)
* LVEF < 25%
* renal failure
* hepatic failure
* known sensitivity to Botulinum toxin
* debilitating neuromuscular disease
* preoperative need for inotropes/vasopressors or intra-aortic balloon pump
* planned MAZE procedure
* history of catheter ablation for AF
* use of Vaughan-Williams class I or III drugs within 5 elimination half lives (or within 2 months for amiodarone)
* undergoing minimally-invasive cardiac surgery
* prior cardiac surgery

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Oh S, Choi EK, Zhang Y, Mazgalev TN. Botulinum toxin injection in epicardial autonomic ganglia temporarily suppresses vagally mediated atrial fibrillation. Circ Arrhythm Electrophysiol. 2011 Aug;4(4):560-5. doi: 10.1161/CIRCEP.111.961854. Epub 2011 Jun 9. PMID 21659633
- [Background] Pokushalov E, Kozlov B, Romanov A, Strelnikov A, Bayramova S, Sergeevichev D, Bogachev-Prokophiev A, Zheleznev S, Shipulin V, Salakhutdinov N, Lomivorotov VV, Karaskov A, Po SS, Steinberg JS. Botulinum toxin injection in epicardial fat pads can prevent recurrences of atrial fibrillation after cardiac surgery: results of a randomized pilot study. J Am Coll Cardiol. 2014 Aug 12;64(6):628-9. doi: 10.1016/j.jacc.2014.04.062. No abstract available. PMID 25104535

RESULTS

PARTICIPANT FLOW:
Groups:
- Epicardial Placebo: After instituting cardiopulmonary bypass (CPB), placebo (normal saline) injections will be performed by the surgeon as follows: Using a standard sterile insulin syringe with a 27g needle, surgeons will inject each of the epicardial fat pads with 1mL of normal saline. After completion of surgery and separation from CPB, patients will proceed along the institutional Cardiac Surgical Caremap. All patients will be monitored with continuous ECG (telemetry) until hospital discharge. POAF will be diagnosed by telemetry or 12-lead ECG, and will be defined as new-onset if it occurs postoperatively at any time before hospital discharge.
  Placebo
Period: Overall Study
Arm/Group | Epicardial Botulinum | Epicardial Placebo
Started | 63 | 67
Completed | 63 | 67
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epicardial Botulinum | Epicardial Placebo | Total
Number analyzed (Participants) | 63 | 67 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (8.6) | 67.5 (9.1) | 67.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 23 | 40
  Male | 46 | 44 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 61 | 67 | 128
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 55 | 57 | 112
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 63 | 67 | 130

OUTCOME MEASURES:

1. Primary Outcome: Time to In-hospital Post-operative Atrial Fibrillation (POAF)
Description: Patients will be seen on a daily basis and the timing of POAF compared between groups. The occurrence of in-hospital POAF will be tracked throughout the hospitalization (up to two weeks) and the time from surgery to the first and subsequent episodes of POAF recorded and compared between groups. POAF will be determined by ECG or telemetry.
Time Frame: From the time of ICU arrival until the time of first documented POAF, or discharge whichever came first, assessed up to 2 weeks
Measure: Mean (Standard Error); unit: hours
Arm/Group | Epicardial Botulinum | Epicardial Placebo
Number analyzed (Participants) | 63 | 67
hours | 224.38 (19.31) | 194.76 (18.36)
Statistical Analysis 1: Comparison: Epicardial Botulinum vs Epicardial Placebo; Test type: Other; p = 0.18, Regression, Cox; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.41 to 1.19]

2. Secondary Outcome: Number of Participants With In-hospital POAF
Description: Patients will be seen on a daily basis and the occurrence of POAF compared between groups.
Time Frame: The incidence of in-hospital POAF will be tracked throughout the hospitalization (up to two weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Epicardial Botulinum | Epicardial Placebo
Number analyzed (Participants) | 63 | 67
Participants | 23 | 32
Statistical Analysis 1: Comparison: Epicardial Botulinum vs Epicardial Placebo; Test type: Other; p = 0.19, Regression, Logistic; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.31 to 1.27]

3. Secondary Outcome: Length of Stay
Description: Total and ICU length of stay will be determined by examining medical records for the length of inpatient hospitalization, assessed over the entire study period (up to two years). ICU and hospital LOS will be recorded and compared between groups
Time Frame: ICU length of stay was measured from time of surgery to time of ICU discharge. Post-operative length of stay was measured from time of surgery to time of hospital discharge.
Measure: Median (Inter-Quartile Range); unit: time in hours
Arm/Group | Epicardial Botulinum | Epicardial Placebo
Number analyzed (Participants) | 63 | 67
time in hours
  ICU LOS in hours | 25.7 [22.4 to 40.2] | 23.1 [20.0 to 34.0]
  Post-operative LOS in hours | 145 [121 to 201] | 149 [125 to 213]
Statistical Analysis 1: Comparison: Epicardial Botulinum vs Epicardial Placebo; ICU length of stay hours; Test type: Other; p = .16, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Epicardial Botulinum vs Epicardial Placebo; Hospital LOS; Test type: Other; p = .51, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Participants With Adverse Events
Description: The total number of postoperative complications (including infectious, neurologic, and renal complications, as well as mortality) and the number of subjects with complications will be monitored and compared between groups.
Time Frame: Adverse events from the time of surgery through hospital discharge, up to 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Epicardial Botulinum | Epicardial Placebo
Number analyzed (Participants) | 63 | 67
Participants | 44 | 47
Statistical Analysis 1: Comparison: Epicardial Botulinum vs Epicardial Placebo; Test type: Other; p = .97, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events from the time of randomization through hospital discharge following study surgery.
Arm/Group | Epicardial Botulinum | Epicardial Placebo
All-Cause Mortality (participants affected / at risk) | 1/63 | 1/67
Serious Adverse Events (participants affected / at risk) | 27/63 | 30/67
Other Adverse Events (participants affected / at risk) | 10/63 | 14/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epicardial Botulinum (N=63) | Epicardial Placebo (N=67)
Atrial Dysrhythmia - Atrial Fibrillation (Cardiac disorders) | 18 | 21
Acute Kidney Injury (Renal and urinary disorders) | 2 | 4
Leukocytosis (Blood and lymphatic system disorders) | 3 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 5
Urinary Tract Infection (Renal and urinary disorders) | 1 | 3
Heart Block (Cardiac disorders) | 1 | 2
Hypotension (Cardiac disorders) | 1 | 2
Ileus (Gastrointestinal disorders) | 1 | 2
Reexploration For Bleeding (Surgical and medical procedures) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Left pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal dysphagia (Nervous system disorders) | 1 | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sternal Wound Infection (Infections and infestations) | 0 | 1
Acute abdomen dilation (Gastrointestinal disorders) | 0 | 1
Acute respiratory failure/hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Altered Mental Status (Nervous system disorders) | 0 | 1
Bilateral Toe and Index finger ischemia. (Vascular disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Dialysis (Renal and urinary disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolemia (Cardiac disorders) | 0 | 1
IABP placement (Cardiac disorders) | 0 | 0
Nausea/Vomiting/Constipation (Gastrointestinal disorders) | 0 | 1
Pacemaker Placement (Cardiac disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Reintubation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Renal Insufficiency (Renal and urinary disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Right sided weakness (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Urinary Incontinence leading to foley re-insertion (Renal and urinary disorders) | 0 | 1
Ventricular Dysrhythmia - Ventricular Tachycardia (Cardiac disorders) | 0 | 1
junctional rhythm (Cardiac disorders) | 1 | 0
post-op hemorrhage, back to OR for re-exploration (Surgical and medical procedures) | 1 | 0
Post-op blood loss anemia requiring transfusions (Blood and lymphatic system disorders) | 0 | 3
prolonged hospitalization c/o coagulation. (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epicardial Botulinum (N=63) | Epicardial Placebo (N=67)
Atrial Dysrhythmia - Atrial Fibrillation (Cardiac disorders) | 5 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT02498769/Prot_SAP_000.pdf